CLINICAL TRIAL: NCT06317428
Title: Change in Serum Levels of NT-proBNP During Triple Therapy With Formoterol/Glycopyrrolate/Budesonide in Patients With COPD.
Brief Title: NT-proBNP Levels During Triple Therapy With Formoterol/Glycopyrrolate/Budesonide in Patients With COPD.
Acronym: NTproBNP
Status: Recruiting | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_001_2024
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: COPD
Keywords: COPD; Formoterol; glycopyrrolate; budesonide; NT-pro-BNP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational prospective study to evaluate serum NT-proBNP levels in a population of COPD patients three months after the iniation of triple inhaled formoterol/glycopyrrolate/budesonide therapy.

DETAILED DESCRIPTION:
The purpose of the trixeo study is to conduct a prospective observational study to evaluate serum NT-proBNP levels in a population of COPD patients three months after the initiation of triple inhaled formoterol/glycopyrrolate/budesonide therapy.

ELIGIBILITY:
Inclusion Criteria:

* COPD;
* Clinical indication for triple inhalation therapy with formoterol/glycopyrrolate/budesonide;

Exclusion Criteria:

* Life expectancy less than one year;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with COPD with clinical indication for triple inhalation therapy with formoterol/glycopyrrolate/budesonide;
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum NT-pro-BNP levels | Before and 3 months after the start of triple therapy with formoterol/glycopyrrolate/budesonide
  Before and 3 months after the introduction of bronchodilator therapy with formoterol/glycopyrrolate/budesonide, patients will be evaluated to assess serum NT-proBNP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Spannella, Study Chair — IRCCS INRCA, Ancona, Italy
Locations (2):
- Italy (2):
  - INRCA Hospital, Ancona
  - IRCCS INRCA Hospital, Osimo